CLINICAL TRIAL: NCT00877214
Title: Prospective Randomized Multicenter Study in First-line Treatment of Advanced progredIeNT Follicular And Other IndoleNt and Mantle Cell Lymphomas
Brief Title: Significance of Duration of Maintenance Therapy With Rituximab in Non-Hodgkin Lymphomas
Acronym: MAINTAIN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jurgen Barth (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor-Investigator, Jurgen Barth, Professor Mathias Rummel, University of Giessen
Organization: University of Giessen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NHL 7-2008
Record Dates: First submitted 2009-04-06; First posted 2009-04-07 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Follicular Lymphomas; Immunocytomas; Marginal Zone Lymphomas; Mantle-Cell Lymphomas; Lymphocytic Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Bendamustine; Rituximab; Significance of maintenance therapy; Efficacy and safety
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — Rituximab; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab (Experimental): Follicular Lymphomas: Rituximab 375 mg/m² for additional 2 years after 2 years of standard maintainance All other lymphomas: Rituximab 375 mg/m² for 2 years as maintainance. From 2014 only Morbus Waldenstroem: Rituximab 1.400 mg absolute s. c. injection
  Interventions: Drug: Rituximab
- Standard (Active Comparator): Rituximab / Observation
  Interventions: Drug: Rituximab / observation

INTERVENTIONS:
Drug: Rituximab — Follicular Lymphomas: induction therapy with bendamustine + rituximab. If CR or PR: Maintenance therapy with rituximab every 2 months for 4 years Immunocytomas, marginal zone and mantle cell lymphomas: induction therapy with bendamustine + rituximab If CR or PR: Maintenance therapy with rituximab every 2 months for 2 years
  Other Names: Mabthera(R); Rituxan(R)
  Arms: Rituximab
Drug: Rituximab / observation — Follicular Lymphomas:induction therapy with bendamustine + rituximab If CR or PR: Maintenance therapy with rituximab every 2 months for 2 years (standard) Immunocytomas, marginal zone and mantle cell lymphomas: induction therapy with bendamustine + rituximab If CR or PR: observation (standard)
  Other Names: Mabthera(R); Rituxan(R)
  Arms: Standard

SUMMARY:
The purpose of this study is to determine if an extended maintenance therapy with Rituximab in follicular and a maintenance therapy in other indolent and mantle cell lymphomas has advantages compared to a shorter or no maintenance therapy.

DETAILED DESCRIPTION:
Results from several randomised studies show a clinical benefit of a maintenance therapy with rituximab in follicular lymphomas. The advantage of a maintenance therapy in other indolent and mantle cell lymphomas is - due to the lower incidence of these diseases- not well investigated.

This study tries to determine the significance of an extended maintenance therapy with rituximab in follicular lymphomas and the significance of a maintenance therapy other indolent and mantle cell lymphomas compared to observation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological verified CD20-positive B-Cell-Lymphoma of the following entities:

  * Follicular Lymphoma Grade 1 and 2
  * Lymphoplasmocytic lymphoma / Immunocytoma (Morbus Waldenström) and small cell lymphocytic lymphoma (CLL without leukemic hemogram)
  * Marginal zone lymphoma, nodal and extra nodal
  * Mantle cell lymphoma
* No prior therapy with cytotoxics, interferon or monoclonal antibodies
* Need for therapy, except mantle cell lymphomas
* Stadium III or IV or Stadium with II bulky disease (> 7 cm diameter, or 3 lesions > 5 cm)
* General condition WHO 0-2
* Age min. 18 years, max. 80 years
* Negative pregnancy test, contraceptives mandatory for women of child-bearing age
* Actual histology, not older than 6 months required
* Written informed consent

Exclusion Criteria:

* Patients not meeting the inclusion criteria above
* Possibility of a primary radiation therapy with curative intention
* Pretreatment, except a single, localized radiation therapy (radiation field not larger than 2 adjacent lymph node regions)
* Co-morbidities, excluding a therapy according to the protocol:

  * severe, medicinal not adjustable hypertension
  * severe limited capacity of the heart (NYHA III or IV), the lung (WHO-Grade III or IV), the liver and kidneys (creatinin > 2 mg/dl, GOT and GPT or bilirubin 3 x ULN), except if caused by lymphoma
  * severe, medicinal not adjustable diabetes mellitus
  * active autoimmune disease
  * active infection, requiring antibiotic therapy
* Patients with proven HIV-infection
* Active replicating hepatitis-Infection
* Severe psychiatric diseases
* Lacking or anticipated non-compliance
* Known hypersensitivity against the active components or additives or mouse- proteins
* Pregnant or nursing women
* Patients with a secondary malignancy or malignant disease in his history if, curative surgery can not be doubtless assured .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1272 (Actual)
Dates: Start 2009-04-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years and ongoing
  Time from randomization until progress or death of any course

SECONDARY OUTCOMES:
Remission rate and duration; event free-, progression free-, disease free- and over all survival | 5 years and ongoing
  Time from randomization until treatment failure due to progression or not achieving any remission; time from achievin CR or PR until progression or relapse

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Rummel, Dr, Principal Investigator — University of Giessen
Locations (1):
- StiL Head Office; Justus-Liebig-University, Giessen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rummel MJ et al. Bendamustin-Rituximab Induction Followed by Observation or Rituximab Maintenance for Newly Diagnosed Patients with Waldenström's Macroglobulinemia: Results From a Prospective, Randomized, Multicenter Study (StiL NHL 7-2008 -MAINTAIN-; ClinicalTrials.gov Identifier: NCT00877214). Blood 2012; 120: 2739. https://doi.org/10.1182/blood.V120.21.2739.2739
- [Background] Immunochemotherapy with Bendamustine-Rituximab (BR) as induction therapy for indolent lymphomas results in a severe lymphopenia with low CD4+ and CD8+ counts without an increase in atypical infections. First results of the infectious disease (ID) project of a prospective, randomized, multicentre study (StiL NHL 7-2008, MAINTAIN; NCT00877214). Hematol Oncol 2013; 31 (Suppl. 1): 106 https://onlinelibrary.wiley.com/doi/pdf/10.1002/hon.2057
- [Background] Rummel MJ et al. Two years rituximab maintenance vs. observation after first-line treatment with bendamustine plus rituximab (B-R) in patients with mantle cell lymphoma: First results of a prospective, randomized, multicenter phase II study (a subgroup study of the StiL NHL7-2008 MAINTAIN trial). DOI: 10.1200/JCO.2016.34.15_suppl.7503 Journal of Clinical Oncology 34, no. 15_suppl (May 2016) 7503-7503.
- [Background] Rummel MJ, et al. Four Versus Two Years of Rituximab Maintenance (R-maintenance) Following Bendamustine Plus Rituximab (B-R): Initial Results of a Prospective, Randomized Multicenter Phase 3 Study in First-Line Follicular Lymphoma (the StiL NHL7-2008 MAINTAIN study). Blood (2017) 130 (Supplement 1): 483.
- [Background] Rummel MJ et al. Two years rituximab maintenance vs. observation after first line treatment with bendamustine plus rituximab (B-R) in patients with marginal zone lymphoma (MZL): Results of a prospective, randomized, multicenter phase 2 study (the StiL NHL7-2008 MAINTAIN trial). DOI: 10.1200/JCO.2018.36.15_suppl.7515 Journal of Clinical Oncology 36, no. 15_suppl (May 20 2018) 7515-7515
- [Background] Rummel MJ et al. Two years Rituximab maintenance vs. observation after first line treatment with Bendamustine plus Rituximab in patients with Marginal Zone Lymphoma (MZL): results from the StiL NHL7-2008 MAINTAIN trial Results of a prospective, randomized, multicentre phase 2 study (a subgroup study of the StiL NHL7-2008 MAINTAIN trial).
- [Background] Rummel MJ et al. Two Years Rituximab Maintenance Vs. Observation after First Line Treatment with Bendamustine Plus Rituximab (B-R) in Patients with Waldenström's Macroglobulinemia (MW): Results of a Prospective, Randomized, Multicenter Phase 3 Study (the StiL NHL7-2008 MAINTAIN trial). Blood (2019) 134 (Supplement_1): 343. https://doi.org/10.1182/blood-2019-121909